CLINICAL TRIAL: NCT02719548
Title: Impact of Breast Shield Designs on Dynamics of Breast Pumping
Acronym: BSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medela AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MBF1505
Record Dates: First submitted 2016-02-12; First posted 2016-03-25 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2016-04

CONDITIONS: Lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Breastshield treatment group A (Experimental): Participants will be treated with the following three breast shields:
  Soft edge oval - Hard oval - Modified PF breast shield Treatment order is described in the corresponding Intervention. Participant will use each breastshield for 2 min after milk ejection.
  Interventions: Device: Soft edge oval - Hard oval - Modified PF breast shield
- Breastshield treatment group B (Experimental): Participants will be treated with the following three breast shields:
  Modified PF breast shield - Soft edge oval - Hard oval Treatment order is described in the corresponding Intervention. Participant will use each breastshield for 2 min after milk ejection.
  Interventions: Device: Modified PF breast shield - Soft edge oval - Hard oval
- Breastshield treatment group C (Experimental): Participants will be treated with the following three breast shields:
  Hard oval - Soft edge oval - Modified PF breast shield Treatment order is described in the corresponding Intervention. Participant will use each breastshield for 2 min after milk ejection.
  Interventions: Device: Hard oval - Soft edge oval - Modified PF breast shield

INTERVENTIONS:
Device: Soft edge oval - Hard oval - Modified PF breast shield — Treatment order:
  1. soft-edge oval breast shield
  2. Hard oval breast shield
  3. modified PersonalFit breast shield
  Other Names: Group A
  Arms: Breastshield treatment group A
Device: Modified PF breast shield - Soft edge oval - Hard oval — 1. modified PersonalFit breast shield
  2. soft-edge oval breast shield
  3. Hard oval breast shield
  Other Names: Group B
  Arms: Breastshield treatment group B
Device: Hard oval - Soft edge oval - Modified PF breast shield — 1. Hard oval breast shield
  2. soft-edge oval breast shield
  3. modified PersonalFit breast shield
  Other Names: Group C
  Arms: Breastshield treatment group C

SUMMARY:
A prospective, randomized, 2-phase/crossover, single center premarket feasibility study. In phase I the comfort will be assessed, the occurence and types of adverse events will be recorded and the assessment how and if the different breast shield designs interact with the lacting breast during pumping. Phase II takes place at home; assessment of adverse events will be recorded and the assessment how the subjects perceives the comfort of the soft edge breast shield during mid term use at home.

DETAILED DESCRIPTION:
This is a prospective, randomized, 2 phase/crossover, single center premarket feasibility study enrolling a total of 15 subjects. Follow up visit will be after 14 days.

The study will be divided in two phases.

The objectives of phase 1 are:

* assessment of Comfort (subjective)
* occurrence and types of adverse events
* to assess if and how the different designs (shapes and soft edge) of the three provided breast shields interacts with the lactating breast during pumping, with regards to:
* The influence of nipple size, diameter and length (measured before pumping)
* Maximum comfortable vacuum selected by participant (mmHg)
* Actual vacuum generated in the tunnel of the breast shields in relation to the vacuum level indicator of the breast pump (mmHg)
* Characteristics of nipple movement in the tunnel during pumping
* Amount of tissue entering the tunnel at maximum applied vacuum (mm)
* Amount of tissue entering the tunnel at minimum applied vacuum (mm)
* Space between breast and shield (mm)

The objectives of phase 2 are

* to assess how the participants perceive the comfort of the soft-edge breast shield during mid term use at home
* to assess which adverse events occur

Study procedures - Phase 1 The participant will be invited for a pumping session (3 times 2 minutes of expression) at Medela Headquarters. The CE-marked Freestyle breast pump and its pumpset will be used in the both phases of the study.The participants will be asked to pump 3 times with each of the 3 breast shields in a randomized order. Each pump session (defined as pump start till pump stop) will be short (2 minutes of pumping after milk ejection has occurred), and all three short pumping session will be done on the left side only. All pump session will start with the stimulation mode and change to expression mode as soon as milk flows.

Study procedures - Phase 2 Once the debriefing is finished the participants will be instructed about the Phase 2 (home use) part of the study and its equipment to be used. Study subjects that do not have a Freestyle system in use, a system will be provided. All subjects will be provided with the applicable breast shield types and introduced as well as the new shields will be handed over.

* the soft-edge breast shield (non CE-marked) and
* the modified PersonalFit Breast Shield (non CE-marked) This part will start for each participant the day after the phase 1assessment at Medela Headquarters.

Day 1-7 (Evaluation of pumping experience with the modified PersonalFit breast shield) Day 7 (Comfort evaluation of the modified PersonalFit breast shield) Day 8-14 (Evaluation of pumping experience with the soft-edge breast shield) Day 14 (Comfort evaluation of the soft-edge breast shield)

ELIGIBILITY:
Inclusion Criteria:

* Female over 18 years
* The participant agrees to pump or feed the last time a minimum of 3 hours before the start of the pumping sessions (phase 1)
* The participant agrees to photograph and video record the breast and upper body (no face) as well as to take audio data.
* Participant agrees to the presence of up to 3 men in the room during the pumping session
* The participant has been pumping at least 7 times in the week prior to study participation, no matter which electric pumps.
* The participant has been consistently pumping 10 ml of milk or more per breast, per pumping session prior to study participation.
* The participant currently use a breast shield size of 24 mm
* The participant has agreed to pump at least 7 times a week over the next three weeks

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Endpoint Phase 1_Optical analysis via photo: pumping sessions of the nipple and breast will be video recorded from the lateral side view; study set up will be filmed and the audio data taken to document all the information | End of phase I (is defined from the date when moms are coming for Phase I, which takes up to 2 weeks. But the visit itself per mom takes approx. 2hours)
  During all three short pumping sessions the nipple and breast will be video recorded from the lateral side view. The study set up will be filmed and the audio data taken to document all the information e.g. nipple movement in the tunnel.
Endpoint Phase 1_Retrospective analysis via Video: by changing the shape of the breast shield the form of the breast shield will better suit and conform to the breast shape | End of phase I (is defined from the date when moms are coming for Phase I, which takes up to 2 weeks. But the visit itself per mom takes approx. 2hours)
  It is theorized that by changing the shape of the breast shield the form of the breast shield will better suit and conform to the breast shape, improving comfort, reducing any point compression against the skin surface, and supporting freedom of movement of the nipple in the tunnel.
  During all three short pumping sessions the nipple and breast will be video recorded from the lateral side view. The study set up will be filmed and the audio data taken to document all the information e.g. nipple movement in the tunnel.
  Retrospective analysis will be undertaken of the recorded videos. The videos will be analyzed using software for a Desktop Ruler. Characteristics of nipple movement in the tunnel during pumping/Amount of tissue entering the tunnel at max.applied vacuum(mm)/Amount of tissue entering the tunnel at min.applied vacuum(mm)/Space between breast and shield(mm)
Endpoint Phase 1_ Questionnaire: After pumping with all 3 breast shields participants will be asked questions about comfort perception, handling experience and the sensation per shield. | End of phase I (is defined from the date when moms are coming for Phase I, which takes up to 2 weeks. But the visit itself per mom takes approx. 2hours)
  After pumping with all 3 breast shields participants will be asked questions about comfort perception, handling experience and the sensation per shield.

SECONDARY OUTCOMES:
Endpoint Phase 2_Pump log and questionnaires: will be asked to document each breast milk expression in the pump log.A questionnaire needs to be completed by the end of each week for the used breast shield | End of phase II (Phase II takes place for 2 weeks at moms home; the end is defined as 4 weeks after end of phase I)
  Participants will be asked to document each breast milk expression in the pump log. The final entries can be compared for both shields, e.g. comparison of max.vacuum comfort (mmHg); milk outcome in mm.
  A questionnaire needs to be completed by the end of each week for the used breast shield as well.
Endpoint Phase 2_Collection of AEs, if any: To assess which adverse events occurred during the home-test by completing the AE form | End of phase II (Phase II takes place for 2 weeks at moms home; the end is defined as 4 weeks after end of phase I)
  - To assess which adverse events occurred during the home-test by completing the AE form

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Prime, PhD, Principal Investigator — Medela AG, Lättichstrasse 4b, 6340 Baar
Locations (1):
- Medela AG, Baar, Canton of Zug, Switzerland

IPD SHARING:
Plan to Share IPD: No